CLINICAL TRIAL: NCT00546598
Title: DURALOC® Option Ceramic-on-Ceramic Hip Prosthesis System PMA Post-approval Study
Brief Title: Post-approval Study of the DURALOC® Option Ceramic-on-Ceramic Hip Prosthesis System
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor withdrew PMA
Sponsor: DePuy Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05024
Record Dates: First submitted 2007-10-17; First posted 2007-10-19 (Estimated); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Non-inflammatory Joint Disease; Osteoarthritis; Avascular Necrosis; Congenital Hip Dysplasia; Post-traumatic Arthritis
Keywords: Total hip replacement, Total hip arthroplasty
MeSH Terms: conditions — Osteoarthritis; Osteonecrosis; Hip Dislocation, Congenital | interventions — Arthroplasty, Replacement, Hip; Arthroplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Duraloc Option COC Hip (Other)
  Interventions: Device: Total hip replacement/arthroplasty

INTERVENTIONS:
Device: Total hip replacement/arthroplasty — Hip replacement
  Other Names: DURALOC® Option Ceramic-on-Ceramic Hip system

SUMMARY:
This study is being conducted to gather medium and long-term information regarding the performance and safety of the commercially available DURALOC® Option Ceramic-on-Ceramic Hip Prosthesis System.

DETAILED DESCRIPTION:
This two-phased study on hip arthroplasty consists of a clinical follow-up phase and a clinical outcomes phase.

The DURALOC® Option Ceramic-on-Ceramic Hip Prosthesis System consists of:

1. a modular ceramic bearing insert that secures to a titanium metal alloy DURALOC® Option Acetabular Shell via a taper locking mechanism; and
2. a ceramic femoral head that is attached to a conventional femoral stem to complete the total hip prosthesis device configuration.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature
* Provide informed consent
* Sufficient acetabular and femoral bone stock to seat the prosthesis
* Willing and able to return for follow-up as specified by the study protocol
* Willing and able to complete the hip outcomes questionnaire and quality of life survey (SF12)
* Undergo hip replacement due to non-inflammatory joint disease, including osteoarthritis, avascular necrosis, congenital hip dysplasia or post-traumatic arthritis.

Exclusion Criteria:

* Diagnosis of inflammatory arthritides such as rheumatoid arthritis, juvenile rheumatoid arthritis, psoriatic arthritis, systemic lupus, erythematosis etc.
* Active infections that may spread to other systems such as osteomyelitis, pyogenic infection of the hip joint overt infection, etc.
* Loss of musculature, neuromuscular compromise or vascular deficiency in the affected limb which impedes evaluation.
* Poor bone quality (e.g. osteoporosis) such that there is concern about the ability of inadequate bone stock to support the implant.
* Morbid obesity
* Involvement in high levels of activity or participation in active sports
* Involvement in heavy manual labor employment
* Increased likelihood of falls due to concomitant illnesses or impairment
* Pregnancy, breast-feeding, a prisoner, mentally incompetent, a known alcohol or drug abuser
* Diagnosis of metabolic disorders or receiving systemic pharmacological treatments leading to progressive deterioration of solid bone support for the implant
* Known history of conditions that may interfere with the total hip arthroplasty survival or outcome (e.g. Paget's disease, Charcot's disease)
* Known presence of active metastatic or neoplastic disease
* Known allergic reactions to implant materials (e.g. ceramic, metal)
* Known history of tissue reactions to implant corrosion or implant wear debris
* Disabilities of other joints that impedes evaluation (e.g. knees, ankles)
* Known presence of highly communicable disease or diseases that may limit follow-up (e.g. immunocompromised conditions, hepatitis, active tuberculosis etc.)
* Previous prosthetic hip replacement device (any type including THA, surface replacement arthroplasty, endoprosthesis etc.)

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2014-04-01 (Actual); Study Completion 2014-04-01 (Actual)

PRIMARY OUTCOMES:
Survivorship | 5 years

SECONDARY OUTCOMES:
Study subject SF-12 health survey | 1, 2 ,3, 4 and 5 years
SF-12 Health survey and Subject Outcomes Questionnaire | 6, 7, 8, 9 and 10 years
Hip Function (using Harris Hip Score) | 6 weeks, 6 months and 1, 2, 3, 4, and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dave Whalen, BS, DC, Study Director — DePuy Orthopaedics
Locations (6):
- United States (6):
  - Northside Hospital, Atlanta, Georgia
  - Memorial Hospital, Springfield, Illinois
  - St. John's Hospital, Springfield, Illinois
  - Fairview Hospital, Cleveland, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Flower Hospital, Sylvania, Ohio